CLINICAL TRIAL: NCT02062242
Title: Electrical Stimulation and Vaginal Palpation in the Pelvic Floor Muscles Awareness: a Randomized Controlled Trial
Brief Title: Electrical Stimulation and Vaginal Palpation in Pelvic Floor Muscles Awareness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Elaine Cristine Lemes Mateus de Vasconcelos, PhD student, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEP 211.405
Record Dates: First submitted 2014-02-01; First posted 2014-02-13 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-02

CONDITIONS: Pelvic Floor Disorders
Keywords: Pelvic Floor; Physical Therapy Specialty; Awareness; Electric Stimulation; Palpation
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Transvaginal electrical stimulation (Experimental): Patients treated with transvaginal electrical stimulation.
  Interventions: Other: Transvaginal electrical stimulation
- Palpation (Experimental): Patients treated with vaginal palpation.
  Interventions: Other: Palpation
- Palpation with posterior pelvic tilt (Experimental): Patients treated with vaginal palpation associated with posterior pelvic tilt and contraction of accessory muscles.
  Interventions: Other: Palpation with posterior pelvic tilt
- Control group (Experimental): Patients receive verbal instructions related to the pelvic floor and its contraction.
  Interventions: Other: Control

INTERVENTIONS:
Other: Transvaginal electrical stimulation — The current employed is biphasic and the stimulation parameters are: frequency of 50 Hz, pulse width of 200 microseconds, contraction time (Ton) of 5 seconds and relaxation time (Toff) of 10 seconds. The current intensity is defined according to the tolerance of patient and the total stimulation time is 20 minutes.
  Arms: Transvaginal electrical stimulation
Other: Palpation — The patient is positioned supine with the lower limbs bent and feet flat on the stretcher. The examiner will hold vaginal palpation and to request her the contraction of PFM. It will be requested 3 sets of 10 contractions with a rest period between contractions. There are two minutes a rest period between sets.
  Arms: Palpation
Other: Palpation with posterior pelvic tilt — The patient is positioned supine with the lower limbs bent and feet flat on the stretcher. The examiner will hold vaginal palpation and to request her the contraction of PFM associated with posterior pelvic tilt and contraction of accessory muscles. It will be requested 3 sets of 10 contractions with a rest period between contractions. There are two minutes a rest period between sets.
  Arms: Palpation with posterior pelvic tilt
Other: Control — The patient receive verbal instructions related to the pelvic floor and its contraction.
  Arms: Control group

SUMMARY:
The purpose of this study is to evaluate the effectiveness of transvaginal electrical stimulation, vaginal palpation, and vaginal palpation associated with posterior pelvic tilt and contraction of accessory muscles in the acquisition of ability to contract the pelvic floor muscles (PFM), as well as to evaluate the sexual function of women studied.

DETAILED DESCRIPTION:
Many women does not know to contract the PFM voluntarily favoring the development of disorders such as urinary and fecal incontinence, pelvic organ prolapse and sexual disorders. However there are no studies in the literature that address the application of therapeutic resources available to improve the PFM awareness. The objective of this study is to evaluate the effectiveness of transvaginal electrical stimulation, vaginal palpation, vaginal palpation associated with posterior pelvic tilt and contraction of accessory muscles in the acquisition of ability to contract the PFM, as well as to evaluate the sexual function of women studied. One hundred twenty women with PFM function graded 0 and 1 measured by Oxford Modified Scale will be submitted at random to physical therapy with transvaginal electrical stimulation, vaginal palpation, vaginal palpation associated with posterior pelvic tilt and contraction of accessory muscles (glutes and hip adductors) and the control group who receive verbal instructions related to the pelvic floor and its contraction. For the evaluation of the sexual function will be applied the Female Sexual Function Index (FSFI).

The patients will be assessed by vaginal palpation, perineometry and surface electromyography before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

Women with age greater than or equal 18 years; Women with pelvic floor muscle function graded 0 and 1 measured by Oxford Modified Scale; Women who voluntarily consente to participate in research.

Exclusion Criteria:

Women with associated neurological pathologies; Women with symptoms of vaginal or urinary tract infection; Women with pelvic organs prolapse graded greater than 2; Pregnancy suspected or confirmed; Cognitive deficit that impedes or impair the procedure.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-03; Primary Completion 2014-06 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the PFM awareness | Baseline, two months
  The transvaginal electrical stimulation, vaginal palpation, and vaginal palpation associated with posterior pelvic tilt and contraction of accessory muscles improve the results in the acquisition of contraction capacity of PFM when compared to controls that receive verbal instructions related to the PFM. The improvement will be assessed through the increase of the grade of vaginal palpation measured by Oxford Modified Scale and through the increase of values of the perineometry and surface eletromyography.

SECONDARY OUTCOMES:
Change from baseline in the sexual function | Baseline, two months
  The improvement of PFM awareness will increase the sexual function of the women studied measured by the increase the score index of FSFI.

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Vasconcelos, PhD student, Principal Investigator — USP Ribeirão Preto; Cristine Ferreira, Mastermind, Study Director — USP Ribeirão Preto
Locations (1):
- Clinical Hospital of Faculty of Medicine of Ribeirão Preto, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Result] Laycock J. Pelvic muscle exercises: physiotherapy for the pelvic floor. Urol Nurs. 1994 Sep;14(3):136-40. No abstract available. PMID 7732416
- [Result] Bo K. Pelvic floor muscle strength and response to pelvic floor muscle training for stress urinary incontinence. Neurourol Urodyn. 2003;22(7):654-8. doi: 10.1002/nau.10153. PMID 14595609
- [Derived] Mateus-Vasconcelos ECL, Brito LGO, Driusso P, Silva TD, Antonio FI, Ferreira CHJ. Effects of three interventions in facilitating voluntary pelvic floor muscle contraction in women: a randomized controlled trial. Braz J Phys Ther. 2018 Sep-Oct;22(5):391-399. doi: 10.1016/j.bjpt.2017.12.006. Epub 2018 Feb 3. PMID 29429823